CLINICAL TRIAL: NCT00392184
Title: Partial Breast Irradiation With Multi-Catheter Brachytherapy for pT1-2pN0 Breast Cancer After Breast Conserving Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: German-Austrian APBI Trial
Record Dates: First submitted 2006-10-24; First posted 2006-10-25 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: accelerated partial breast irradiation; multicatheter brachytherapy; high dose rate brachytherapy; pulsed dose rate brachytherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- APBI (Experimental): Accelerated Partial Breast Irradiation with interstitial Brachytherapy
  Interventions: Procedure: Accelerated partial breast irradiation

INTERVENTIONS:
Procedure: Accelerated partial breast irradiation

SUMMARY:
The purpose of this study is to determine whether accelerated partial breast irradiation (APBI) with multi-catheter brachytherapy is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* pT1/2 (≤ 3 cm)
* pN0 or pN1 mi
* M0 and no contralateral BC
* Clear margins (≥ 2 mm)
* Age ≥ 35 years
* ER and/or PR positive

Exclusion Criteria:

* Multifocality or Multicentricity
* EIC
* Lymphovascular invasion
* Poorly differentiated tumors
* Diffuse microcalcifications

Ages: 35 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2000-11; Primary Completion 2009-02 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vratislav Strnad, MD, Study Chair — University Hospital Erlangen, Germany; Oliver J Ott, MD, Study Director — University Hospital Erlangen, Germany; Guido Hildebrandt, MD, Principal Investigator — University Hospital Leipzig, Germany; Richard Pötter, MD, Principal Investigator — University Hospital AKH Vienna, Austria; Joe Hammer, MD, Principal Investigator — Hospital Barmherzige Schwestern Linz, Austria
Locations (4):
- Austria (2):
  - Hospital Barmherzige Schwestern Linz, Linz
  - University Hospital AKH Vienna, Vienna
- Germany (2):
  - University Hospital Erlangen, Erlangen
  - University Hospital Leipzig, Leipzig

REFERENCES:
- [Result] Ott OJ, Potter R, Hammer J, Hildebrandt G, Lotter M, Resch A, Pohls U, Beckmann MW, Sauer R, Strnad V. Accelerated partial breast irradiation with iridium-192 multicatheter PDR/HDR brachytherapy. Preliminary results of the German-Austrian multicenter trial. Strahlenther Onkol. 2004 Oct;180(10):642-9. doi: 10.1007/s00066-004-1294-2. PMID 15480513
- [Result] Strnad V, Ott O, Potter R, Hildebrandt G, Hammer J, Resch A, Lotter M, Ackermann S, Beckmann MW, Sauer R. Interstitial brachytherapy alone after breast conserving surgery: interim results of a German-Austrian multicenter phase II trial. Brachytherapy. 2004;3(3):115-9. doi: 10.1016/j.brachy.2004.08.003. PMID 15533801
- [Result] Ott OJ, Potter R, Hildebrandt G, Hammer J, Lotter M, Beckmann MW, Sauer R, Strnad V. [Partial breast irradiation for early breast cancer with favorable prognostic factors: 3-year results of the German-Austrian phase II-trial]. Rofo. 2005 Jul;177(7):962-7. doi: 10.1055/s-2005-858268. German. PMID 15973598
- [Derived] Ott OJ, Hildebrandt G, Potter R, Hammer J, Hindemith M, Resch A, Spiegl K, Lotter M, Uter W, Kortmann RD, Schrauder M, Beckmann MW, Fietkau R, Strnad V. Accelerated partial breast irradiation with interstitial implants: risk factors associated with increased local recurrence. Int J Radiat Oncol Biol Phys. 2011 Aug 1;80(5):1458-63. doi: 10.1016/j.ijrobp.2010.04.032. Epub 2010 Aug 2. PMID 20675064